CLINICAL TRIAL: NCT03003910
Title: Efficacy of a Positive Psychological Intervention in Patients With Eating Disorders: a Randomized Control Trial
Brief Title: Efficacy of a Positive Psychological Intervention in Patients With Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Hospital Provincial de Castellon (Other); PREVI Clinical Center (Unknown)
Responsible Party: Principal Investigator, Angel Enrique Roig, Ph.D Student, Universitat Jaume I
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aenrique
Record Dates: First submitted 2016-12-19; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Eating Disorder; Daily Activities
Keywords: Best Possible Self
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Activities of Daily Living

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Best Possible Self (Experimental): Participants are asked to write and imagine about a future in which they have reached all their goals and they have developed all their potentialities in four different domains: personal, professional, social and health domain.
  They carry out the exercise in a Positive Technology System called the "Book of Life", which has shown efficacy in the enhancement of positive mood (Baños, Etchemendy, Farfallini, García-Palacios, Quero & Botella, 2014). This application looks like a personal diary, where participants can write all that they want and these essays are supported by multimedia content (pictures, songs and videos). Additionally, they can continue doing the exercise in a web platform in which they can visualize all the content they had developed previously.
  Interventions: Behavioral: Best Possible Self
- Daily Activities (Placebo Comparator): Participants are asked to think and write about all that they have done the last 24 hours. They carry out the exercise in a powerpoint document, where they can record all the activities, situations and thoughts occurred in the past 24 hours.
  Interventions: Behavioral: Daily Activities

INTERVENTIONS:
Behavioral: Best Possible Self — Intervention group which requires people to envision themselves in a future in which all has gone in the best possible way.
  Other Names: Positive Psychological Intervention
  Arms: Best Possible Self
Behavioral: Daily Activities — Control group which consists of thinking and writing about all the activities and situations that had taken place during the last 24 h.
  Arms: Daily Activities

SUMMARY:
This study is aimed to test the efficacy of a positive psychological intervention for promoting positive emotions and optimistic thinking in eating disordered patients. Participants are randomly assigned to receive the positive intervention or the control condition, which consists on thinking about daily activities.

DETAILED DESCRIPTION:
Eating disorders (ED) are very difficult conditions to treat. Therefore, interventions in this field are shifting their main target towards the disorder's impact in quality of life, rather than ED symptomatology in itself. In this sense, a focus in the promotion of positive emotions and well-being is emerging in order to buffer from the harmful effects caused by ED.

Positive psychological interventions have shown efficacy in the promotion of positive emotions and well-being. In this sense, one of these interventions is called Best Possible Self (BPS), since is aimed to enhance positive emotions and well-being. Specifically, BPS is a positive future thinking technique, which requires people to envision themselves in the future, after everything has gone as good as it possibly could. This exercise has shown efficacy improving optimism, future expectancies and positive affect compared to a control condition, in general population and depressive patients.

Furthermore, the progress of Information and Communication Technologies, has allowed the development of technology applications and devices that could enhance the quality of experience and the well-being levels. This approach is called Positive Technology and it can be used as a complement to positive psychological interventions. Positive Technology can be defined as the scientific and applied approach to improve the quality of our personal experience trying to increase wellness and generate strengths.

Taking into account the prior literature, the aim of the present study is to carry out a randomized controlled study with ED patients in order to explore if BPS is able to produce improvements in different well-being and clinical measures. The exercise will be applied through a Positive Technology system. The design employed in this study is similar to the used in other studies.

Five assessment moments were used: Before the exercise (baseline), after the first session (day 1) and post-training (1 month). Moreover, two follow-ups were included: one month after finishing the training period (1st follow-up) and three months after finishing the training (2nd follow-up)

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of Eating Disorder by a Clinical Psychologist according to DSM-IV criteria
* Subject accepts to participate in the study voluntarily

Exclusion Criteria:

* Subject suffering a severe physical condition
* Subject suffering from substance or alcohol depedence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Subjective Probability Task (SPT; MacLeod, 1996). Change assessment. | Baseline, day 1, 1 month, 2 months, 4 months
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 y 0.91, respectively).
Positive and Negative Affect Scale (PANAS, Watson, Clark & Tellegen, 1988; Sandín et al., 1999). Change assessment. | Baseline, day 1, 1 month, 2 months, 4 months
  To measure affect, the Spanish adaptation of the Positive and Negative Affect Scale was used (PANAS, Sandín et al., 1999; Watson, Clark & Tellegen, 1988). This instrument is composed of 20 items: 10 items measuring positive affective states and 10 items measuring negative affect states. Participants rate on a five-point scale (from "Not at all" to "Extremely") the degree to which they usually feel a specific affective state. PANAS is one of the most widely-used instruments to measure affect because it shows excellent psychometric properties (Cronbach Alpha's from 0.87-0.91).

SECONDARY OUTCOMES:
Life Orientation Test (Lot-R; Otero, Luengo, Romero Gómez & Castro, 1998; Scheier, Carver & Bridges, 1994). Change assessment. | Baseline, 1 month, 2 months, 4 months
  This scale measures positive and negative expectancies about future events. It consists of 20 statements referring to negative expectancies and 10 statements referring to positive expectancies. Participants answer on a 7-point scale (Not at all likely to occur - Extremely likely to occur). Some studies have found an appropriate levels of internal consistency for positive and negative expectancies (α=0.80-0.82 y 0.91, respectively).
General Self Efficacy Scale-12 (GSES-12; Bosscher et al., 1997; Herrero et al., 2014). Change assessment. | Baseline, 1 month, 2 months, 4 months
  This questionnaire evaluates a general dimension and three aspects of self-efficacy: initiative, persistence and effort. The internal consistency coefficients for the subscales varied from excellent to good (Initiative = 0.83; Effort =0.77; Persistence = 0.80; and Total = 0.86).
Dispositional Hope Scale (DHS; Snyder et al., 1991). Change assessment. | Baseline, 1 month, 2 months, 4 months
  This instrument evaluates dispositional hope. It is composed of 12 items (Agency: 4 items; Pathways= 4 items; Fillers= 4 items), with an 8-point Likert scale ranging from 1 (definitely false) to 8 (definitely true). Internal consistency coefficient (Cronbach's alpha) for the total scale was excellent (.89).
Self-Concordant Motivation (SCM; Sheldon & Elliot, 1999) | day 1
  This instrument assesses participants' initial motivation to do the assigned exercise. It explores the different reasons for the participants to carry out the exercise. The scale is composed of 4 items whose goal is to find out whether the motivation is intrinsic or extrinsic. A total score is obtained by subtracting the two extrinsic motivation scores from the two intrinsic motivation scores.

OTHER OUTCOMES:
Eysenck Personality Questionnaire - Revised - Neuroticism (EPQ-R-N; Eysenck, Eysenck & Barrett, 1985; Eysenck & Eysenck, 1997). | Baseline
  This scale assesses the neuroticism level of the individual, showing if he is stable or neurotic. This subscale is composed by 12 items of dicotomic response (yes-not). Regarding psychometric properties, Eysenck and Eysenck (1997) got an alpha coefficient between 0-73 and 0.82.
Eating Attitudes Test (EAT-26; Garner, Olmsted, Bohr & Garfinkel, 1982) | Baseline
  This questionnaire assesses a broad range of attitudes and behaviors related to anorexia nervosa. It is composed of 26 items rated on a 6-point Likert scale from 0 (never) to 6 (always), based on the frequency with which the individual carries out the behavior or has the thought described by the item. The instrument has shown excellent psychometric properties (Toro, Castro, Garcia, Perez & Cuesta, 1989; Rivas, Bersabé, Jiménez & Berrocal, 2010).
Brief Symptom Inventory (Ruipérez, Ibañez, Lorente, Moro & Ortet, 2001) | Baseline
  This scale encompass ninve primary dimensions of psychopathological symptoms: psychoticism, somatization, depression, hostility, phobic anxiety, obsessive-compulsive, anxiety (panic), paranoid ideation, and nervous tension. Each BSI item is rated on a 5- point scale (0 to 4) according to manifestations of symptoms in the last 30 days (ranging from "not at-all" to "extremely").

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, Professor, Study Director — University Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bolier L, Haverman M, Kramer J, Westerhof GJ, Riper H, Walburg JA, Boon B, Bohlmeijer E. An Internet-based intervention to promote mental fitness for mildly depressed adults: randomized controlled trial. J Med Internet Res. 2013 Sep 16;15(9):e200. doi: 10.2196/jmir.2603. PMID 24041479
- [Background] Botella C, Riva G, Gaggioli A, Wiederhold BK, Alcaniz M, Banos RM. The present and future of positive technologies. Cyberpsychol Behav Soc Netw. 2012 Feb;15(2):78-84. doi: 10.1089/cyber.2011.0140. Epub 2011 Dec 9. PMID 22149078
- [Background] Meevissen YM, Peters ML, Alberts HJ. Become more optimistic by imagining a best possible self: effects of a two week intervention. J Behav Ther Exp Psychiatry. 2011 Sep;42(3):371-8. doi: 10.1016/j.jbtep.2011.02.012. Epub 2011 Mar 2. PMID 21450262
- [Background] Pietrowsky, R., & Mikutta, J. (2012). Effects of positive psychology interventions in depressive patients-A randomized control study. Psychology, 3(12), 1067. doi: 10.4236/psych.2012.312158.
- [Background] Renner F, Schwarz P, Peters ML, Huibers MJ. Effects of a best-possible-self mental imagery exercise on mood and dysfunctional attitudes. Psychiatry Res. 2014 Jan 30;215(1):105-10. doi: 10.1016/j.psychres.2013.10.033. Epub 2013 Nov 1. PMID 24252218
- [Background] Sheldon, K. M., & Lyubomirsky, S. (2006). How to increase and sustain positive emotion: The effects of expressing gratitude and visualizing best possible selves. The Journal of Positive Psychology, 1(2), 73-82.
- [Background] Dawson L, Rhodes P, Touyz S. "Doing the impossible": the process of recovery from chronic anorexia nervosa. Qual Health Res. 2014 Apr;24(4):494-505. doi: 10.1177/1049732314524029. Epub 2014 Mar 4. PMID 24594747
- [Background] Noordenbos G, Oldenhave A, Muschter J, Terpstra N. Characteristics and treatment of patients with chronic eating disorders. Eat Disord. 2002 Spring;10(1):15-29. doi: 10.1080/106402602753573531. PMID 16864242
- [Background] Tchanturia K, Dapelo MA, Harrison A, Hambrook D. Why study positive emotions in the context of eating disorders? Curr Psychiatry Rep. 2015 Jan;17(1):537. doi: 10.1007/s11920-014-0537-x. PMID 25413641
- [Derived] Enrique A, Breton-Lopez J, Molinari G, Roca P, Llorca G, Guillen V, Fernandez-Aranda F, Banos RM, Botella C. Implementation of a Positive Technology Application in Patients With Eating Disorders: A Pilot Randomized Control Trial. Front Psychol. 2018 Jun 11;9:934. doi: 10.3389/fpsyg.2018.00934. eCollection 2018. PMID 29942272